CLINICAL TRIAL: NCT00072358
Title: Phase II Study of Anti-GD2 3F8 Antibody and GM-CSF for High-Risk Neuroblastoma
Brief Title: Monoclonal Antibody 3F8 and Sargramostim in Treating Patients With Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-077; MSKCC-03077
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma; localized unresectable neuroblastoma; recurrent neuroblastoma; regional neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Population Groups

ARMS (2):
- patients have refractory bone marrow disease (Experimental): This phase II trial of the anti-GD2 murine IgG3 monoclonal antibody 3F8 combined with granulocyte-macrophage colony stimulating factor (GM-CSF) will assess response of minimal residual disease (MRD) in patients with high-risk neuroblastoma (NB) and help establish the optimal way to use GM-CSF.
  Interventions: Biological: anti-GD2 murine IgG3 monoclonal antibody 3F8
- patients have no evidence of disease (Experimental): This phase II trial of the anti-GD2 murine IgG3 monoclonal antibody 3F8 combined with granulocyte-macrophage colony stimulating factor (GM-CSF) will assess response of minimal residual disease (MRD) in patients with high-risk neuroblastoma (NB) and help establish the optimal way to use GM-CSF.
  Interventions: Biological: anti-GD2 murine IgG3 monoclonal antibody 3F8

INTERVENTIONS:
Biological: anti-GD2 murine IgG3 monoclonal antibody 3F8 — The total dosage of 3F8 per cycle is the same as in prior trials (100 mg/m2), administered at 20 mg/m2/day and infused over ~1.5 hr or less (0.5 hr is customary), with analgesics and antihistamines used as needed for expected side-effects. 3F8 is started ~1 hr after completion of GM-CSF administration. GM-CSF is dosed at 250 mcg/m2/day from day -5 to day +1 (Wednesday to Tuesday is customary) , and is 500 mcg/m2/day thereafter (i.e., on days +2 to +4; Wednesday to Friday), as in the predecessor protocol.18,74 Patients come off study if progressive disease occurs or if there is life-threatening grade 4 toxicity from 3F8; otherwise, patients will receive a minimum of 4 cycles of treatment and will continue treatment through 24 months. It is expected that patients will receive ~10 cycles.
  Other Names: patients (enrolled on study for treatment of primary refractory disease), the; break between end of a cycle of 3F8/GM-CSF and start of next cycle is 2-to-4-weeks through 4; cycles after achievement of CR in BM; subsequent breaks are ~8 weeks. In this; group, isotretinoin is started after documentation of response to, and after; >2 cycles of, 3F8/GM-CSF.
  Arms: patients have refractory bone marrow disease
Biological: anti-GD2 murine IgG3 monoclonal antibody 3F8 — The total dosage of 3F8 per cycle is the same as in prior trials (100 mg/m2), administered at 20 mg/m2/day and infused over ~1.5 hr or less (0.5 hr is customary), with analgesics and antihistamines used as needed for expected side-effects. 3F8 is started ~1 hr after completion of GM-CSF administration. GM-CSF is dosed at 250 mcg/m2/day from day -5 to day +1 (Wednesday to Tuesday is customary) , and is 500 mcg/m2/day thereafter (i.e., on days +2 to +4; Wednesday to Friday), as in the predecessor protocol.18,74 Patients come off study if progressive disease occurs or if there is life-threatening grade 4 toxicity from 3F8; otherwise, patients will receive a minimum of 4 cycles of treatment and will continue treatment through 24 months. It is expected that patients will receive ~10 cycles.
  Other Names: For Group 2 patients (enrolled on study in CR/VGPR, i.e., with no evidence of disease),; the break between end of a cycle and start of next cycle is 2-to-4 weeks through 4 cycles;; subsequent breaks are ~8 weeks. Isotretinoin is started after cycle 2 of 3F8/GM-CSF. Road; map/schema is in section 4.2. Regarding patients in second or greater CR from relapse in the; central nervous system, if they develop early HAMA which precludes timely completion of the; minimum of 4 cycles of 3F8/GM-CSF, they are eligible to go off protocol, to be treated with; low-dose maintenance regimens of irinotecan,94 temozolomide,95 or the two agents combined;96; they can resume treatment with 3F8/GM-CSF if HAMA becomes negative.
  Arms: patients have no evidence of disease

SUMMARY:
RATIONALE: Monoclonal antibodies, such as monoclonal antibody 3F8, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Colony-stimulating factors, such as sargramostim, may increase the number of immune cells found in bone marrow or peripheral blood. Combining monoclonal antibody 3F8 with sargramostim may cause a stronger immune response and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining monoclonal antibody 3F8 with sargramostim in treating patients who have neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of sargramostim (GM-CSF) in enhancing monoclonal antibody 3F8-mediated ablation in patients with high-risk neuroblastoma.
* Determine the prognostic impact of minimal residual bone marrow disease on relapse-free survival of patients treated with this regimen.
* Compare the effects of short-term (2-hour intravenous) vs prolonged (subcutaneous release) daily GM-CSF on granulocyte activation, in order to establish the optimal route for tumor-cell kill in these patients.

OUTLINE: This is an open-label study. Patients are stratified according to evaluable disease (yes [primary refractory bone marrow disease] vs no [no evidence of disease]).

Patients receive sargramostim (GM-CSF) subcutaneously on days -5 to 4 and monoclonal antibody 3F8 IV over 0.5-1.5 hours on days 0-4. Treatment repeats every 3 weeks for 4 courses and then every 8 weeks for up to a total of 24 months in the absence of disease progression or unacceptable toxicity.

Beginning after 2 courses of GM-CSF and monoclonal antibody 3F8, patients also receive oral isotretinoin twice daily on days 1-14 (when no monoclonal antibody 3F8 is administered). Treatment with isotretinoin repeats approximately every 28 days for 6 courses.

PROJECTED ACCRUAL: A total of 340 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma by histopathology OR bone marrow metastases and high urine catecholamine levels
* Disease must meet risk-related treatment guidelines and any of the following International Neuroblastoma Staging System stages:

  * Stage 4 with (any age) OR without (> 18 months of age of age) MYCN amplification
  * MYCN-amplified other than stage 1
* No evidence of disease (i.e., in complete response/remission or very good partial response/remission) OR disease resistant to standard therapy (i.e., incomplete response in bone marrow)
* No progressive disease or MIBG-avid soft tissue tumor

PATIENT CHARACTERISTICS:

* No existing renal, cardiac, hepatic, neurologic, pulmonary, or gastrointestinal toxicity ≥ grade 3
* No human anti-mouse antibody (HAMA) titer greater than 1,000 Elisa units/mL
* No history of allergy to mouse proteins
* No active life-threatening infection
* Not pregnant
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2003-07; Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian H. Kushner, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Kushner BH, Modak S, Basu EM, Roberts SS, Kramer K, Cheung NK. Posterior reversible encephalopathy syndrome in neuroblastoma patients receiving anti-GD2 3F8 monoclonal antibody. Cancer. 2013 Aug 1;119(15):2789-95. doi: 10.1002/cncr.28137. Epub 2013 Apr 30. PMID 23633099
- [Derived] Cheung IY, Hsu K, Cheung NK. Activation of peripheral-blood granulocytes is strongly correlated with patient outcome after immunotherapy with anti-GD2 monoclonal antibody and granulocyte-macrophage colony-stimulating factor. J Clin Oncol. 2012 Feb 1;30(4):426-32. doi: 10.1200/JCO.2011.37.6236. Epub 2011 Dec 27. PMID 22203761

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Refractory Bone Marrow Disease and High Risk of Recurrence: Participants included have refractory bone marrow disease and high risk of recurrence of refractory bone marrow disease. All participants will receive anti-GD2 murine IgG3 monoclonal antibody 3F8. As per the study team, the data were not collected in the manner requested. As a result they cannot separate the patients into the respective protocol groups
Period: Overall Study
Arm/Group | Participants With Refractory Bone Marrow Disease and High Risk of Recurrence
Started | 291
Completed | 291
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Participants With Refractory Bone Marrow Disease and High Risk of Recurrence
Number analyzed (Participants) | 291
Age, Continuous [Median (Full Range); unit: years] | 4 [0 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112
  Male | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 270
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 28
  White | 238
  More than one race | 0
  Unknown or Not Reported | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 291

OUTCOME MEASURES:

1. Primary Outcome: Efficacy at Completion of Treatment
Time Frame: 3 years
Population: Data were not collected
Groups:
- Participants With Refractory Bone Marrow Disease and High Risk of Recurrence: Participants included have refractory bone marrow disease and high risk of recurrence of refractory bone marrow disease. All participants will receive anti-GD2 murine IgG3 monoclonal antibody 3F8
Arm/Group | Participants With Refractory Bone Marrow Disease and High Risk of Recurrence
Number analyzed (Participants) | 0

2. Primary Outcome: Relapse-free Survival Every 3 Months
Time Frame: 3 years
Population: Data were not collected
Arm/Group | Participants With Refractory Bone Marrow Disease and High Risk of Recurrence
Number analyzed (Participants) | 0

3. Secondary Outcome: Compare Granulocyte Activation in Patients Treated With Short-term vs Prolonged Daily Exposure to Sargramostim (GM-CSF) After 4 Courses
Time Frame: 3 years
Population: Data were not collected
Arm/Group | Participants With Refractory Bone Marrow Disease and High Risk of Recurrence
Number analyzed (Participants) | 0

4. Secondary Outcome: Simplify Treatment With Consequent Reduction in Cost
Time Frame: 3 years
Population: Data were not collected
Arm/Group | Participants With Refractory Bone Marrow Disease and High Risk of Recurrence
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Participants With Refractory Bone Marrow Disease and High Risk of Recurrence
All-Cause Mortality (participants affected / at risk) | 135/291
Serious Adverse Events (participants affected / at risk) | 153/291
Other Adverse Events (participants affected / at risk) | 287/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Refractory Bone Marrow Disease and High Risk of Recurrence (N=291)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1
Allergic Reaction/Hyper (Immune system disorders) | 11
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Ataxia (Nervous system disorders) | 1
Blood,Bone marrow,other (Blood and lymphatic system disorders) | 1
CNS hemorrhage (Nervous system disorders) | 2
Cardiac left vent (Cardiac disorders) | 1
Cardiovascular, Arrhythmia other (Cardiac disorders) | 1
Cardiovascular, other (Cardiac disorders) | 2
Catheter-rel inf (Infections and infestations) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Depressed level of cons (Nervous system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 8
Dysphagia, esophagitis (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (General disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 11
Fever (General disorders) | 121
GI, other (Gastrointestinal disorders) | 2
Headache (Nervous system disorders) | 4
Hematemesis (Gastrointestinal disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 9
Hypotension (Vascular disorders) | 10
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9
Infection unk ANC (Infections and infestations) | 6
Infection w.out neutropenia (Infections and infestations) | 57
Infection with grade 3/4 neut (Infections and infestations) | 3
Infection/Feb Neut-Other (Infections and infestations) | 1
Irritability < 3 years (Psychiatric disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 2
Middle ear/hearing (Ear and labyrinth disorders) | 2
Mood alteration-anxiety (Psychiatric disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Neurology, other (Nervous system disorders) | 6
Neutrophils/gran (Investigations) | 5
Pain, other (General disorders) | 5
Platelets (Investigations) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 1
Rash, desquamation (Skin and subcutaneous tissue disorders) | 2
Rigors, chills (General disorders) | 18
SGPT (ALT) (Investigations) | 3
Secondary malignancy, other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Seizure (Nervous system disorders) | 4
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 9
Thrombosis (Vascular disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Vomiting (Gastrointestinal disorders) | 16
Weight loss (Investigations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Refractory Bone Marrow Disease and High Risk of Recurrence (N=291)
Pain, other (General disorders) | 157
Urticaria (Skin and subcutaneous tissue disorders) | 142
Flushing (Vascular disorders) | 103
Pruritus (Skin and subcutaneous tissue disorders) | 100
Vomiting (Gastrointestinal disorders) | 90
Cough (Respiratory, thoracic and mediastinal disorders) | 80
Nausea (Gastrointestinal disorders) | 78
Fever (General disorders) | 63
Edema (General disorders) | 58
Dry skin (Skin and subcutaneous tissue disorders) | 53
Rash, desquamation (Skin and subcutaneous tissue disorders) | 42
Headache (Nervous system disorders) | 40
Diarrhea (Pts w/out col) (Gastrointestinal disorders) | 38
Anorexia (Metabolism and nutrition disorders) | 35
Injection site reaction (General disorders) | 33
Pulmonary, other (Reproductive system and breast disorders) | 32
Bone pain (Musculoskeletal and connective tissue disorders) | 29
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 24
Mood alteration-anxiety (Psychiatric disorders) | 22
Abdominal pain/cramping (Gastrointestinal disorders) | 20
Constipation (Gastrointestinal disorders) | 19
Fatigue (General disorders) | 18
Hypertension (Vascular disorders) | 18
Allergy, other (Immune system disorders) | 16
Hypotension (Vascular disorders) | 16
Irritability < 3 years (Psychiatric disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT00072358/Prot_SAP_000.pdf